CLINICAL TRIAL: NCT00128154
Title: A Double-Blind Randomized Controlled Clinical Trial of Chromium Picolinate on Clinical and Biochemical Features of the Metabolic Syndrome
Brief Title: Chromium Picolinate for the Treatment of Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21 AT001147-01
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Metabolic Syndrome X; Prediabetic State; Insulin Resistance; Obesity; Metabolic Diseases
Keywords: Chromium; Chromium picolinate; Blood Glucose; Cholesterol; Complementary Therapies
MeSH Terms: conditions — Metabolic Syndrome; Prediabetic State; Insulin Resistance; Obesity; Metabolic Diseases | interventions — picolinic acid

INTERVENTIONS:
Drug: Chromium picolinate

SUMMARY:
The purpose of this study is to determine whether chromium supplements can reduce symptoms of metabolic syndrome, a collection of symptoms that increase one's risk for developing heart disease, stroke, and diabetes.

DETAILED DESCRIPTION:
Metabolic syndrome is a serious condition that may lead to a number of life-threatening diseases. A reduction in the symptoms of metabolic syndrome could result in decreased morbidity and health care costs and increased quality of life.

Chromium is an essential mineral that is used in the breakdown of fats, protein, and carbohydrates. The cholesterol-lowering and blood sugar-stabilizing properties of chromium make the supplement a strong candidate for reducing the symptoms of metabolic syndrome. This study will determine whether chromium supplements can reduce symptoms of metabolic syndrome in abdominally obese individuals.

Participants will be randomly assigned to receive either chromium supplements or placebo daily for 16 weeks. Participants will have study visits at study start and at Months 2 and 4. A follow-up visit will occur 5 months after the end of the intervention period. Blood tests, urine tests, and nail clippings will be used to assess lipoprotein cholesterol, insulin response to glucose, lean body mass, blood pressure, oxidative stress, and chromium levels in participants.

ELIGIBILITY:
Inclusion Criteria:

* Meet at least two of the following criteria for diagnosis of metabolic syndrome: 1) systolic blood pressure higher than 130 mmHg or diastolic blood pressure higher than 85 mmHg in untreated patients OR use of more than one approved antihypertensive agent; 2) fasting glucose higher than 110 mg/dL; 3) fasting triglycerides higher than 150 mg/dL; 4) high density lipoprotein (HDL) less than 40 mg/dL for men and less than 50 mg/dL for women
* Abdominal obesity defined by a waist circumference higher than 40 inches for men and 35 inches for women

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Use of antihyperglycemic or insulin sensitizing medication within 3 months prior to study entry
* Uncontrolled hypertension
* Triglycerides higher than 800 mg/dL
* Low density lipoprotein (LDL) cholesterol higher than 190 mg/dL
* History of renal insufficiency
* History of liver disease or abnormal liver function tests (higher than 3x upper limit normal)
* History of atherosclerotic cardiovascular disease
* History of congestive heart failure
* Cancer within 5 years prior to study entry. Participants with a history of skin cancer are not excluded.
* Surgery within 30 days prior to study entry
* Use of niacin within 6 weeks prior to study entry
* Use of fibrates within 12 weeks prior to study entry
* History of alcohol or drug abuse
* Participation in an investigational drug study within 6 weeks prior to study entry
* Any major active rheumatologic, pulmonary, or dermatologic disease, or inflammatory condition
* Unstable medical or psychological condition that would interfere with the study
* Use of any chromium-containing dietary supplement within 3 months prior to study entry
* Allergy or sensitivity to chromium, picolinic acid, or chromium picolinate
* Use of beta blockers, corticosteroids, androgens, anticoagulants, and antiarrhythmics within 3 months prior to study entry
* Use of dietary supplements within 30 days prior to study entry. Participants who use multivitamins, calcium, vitamin D, or (non-niacin) B vitamins are not excluded.
* Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-01; Study Completion 2005-12

PRIMARY OUTCOMES:
Increase in insulin sensitivity

SECONDARY OUTCOMES:
Glucose effectiveness
acute insulin response to glucose
fasting triglycerides and high density lipoprotein cholesterol
free fatty acids
weight and/or body composition

CONTACTS AND LOCATIONS:
Overall Officials: Nayyar Iqbal, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Iqbal N, Cardillo S, Volger S, Bloedon LT, Anderson RA, Boston R, Szapary PO. Chromium picolinate does not improve key features of metabolic syndrome in obese nondiabetic adults. Metab Syndr Relat Disord. 2009 Apr;7(2):143-50. doi: 10.1089/met.2008.0048. PMID 19422140